CLINICAL TRIAL: NCT06465212
Title: Personalized Shared Eye-care Identification of Age-related Macular Degeneration Using Artificial Intelligence and Telemedicine in a Prospective, Exploratory, Multinational, Multicentre Cross-sectional Study Matching Optometrist Office-based Sites With Clinical Supervision
Brief Title: Personalized Shared Eye-care Identification of Age-related Macular Degeneration Using Artificial Intelligence and Telemedicine by Matching Optometrist Office-based Sites With Clinical Supervision
Acronym: PYRENEES
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ursula Schmidt-Erfurth, M.D., Prof., Medical University of Vienna
Other Study IDs: 1318/2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Age-Related Macular Degeneration
Keywords: Telemedicine; Ophthalmic Coherence Tomography; Shared-care
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TopCon Maestro 2 OCT — Ophthalmic Coherence Tomography

SUMMARY:
Office-based optometrist centres equipped with low-cost OCT devices can be used for screening of age-related macular degeneration. Matching next-door optometrist centres with clinical sites introduces a shared care service in an unprecedented and broad manner and offers timely and inclusive access to eye care for all citizens affected by the most frequent blinding disease in western countries.

The aim of the study is to detect AMD in a next-door office-based setting on an individual level using low-cost OCT, through a telemedicine feedback loop.

The specific aims of this study are:

* Setting up a network of optometrist centres matched to clinical sites to perform shared care to protect eyesight in the elderly population.
* Identify imaging biomarkers of age-related macular degeneration from OCT imaging.
* Give a risk estimation of progression using a one-time low-cost OCT scan

ELIGIBILITY:
Inclusion Criteria:

* Age: 55-99 years old
* Preserved visual function, defined as visual acuity better than or equal to 0.3logMAR in one or both eyes

Exclusion Criteria:

* Refractive errors with mean spherical equivalent (MSE) greater than +/-6.00, with no limit to astigmatic component.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Allcomers at the optometrist office that meet the inclusion criteria. In general, there is no specific targeting in recruitment. This collection of data does not represent a traditional clinical study that is recruiting patients, but is exclusively collecting images from asymptomatic individuals.
  Individuals are imaged within the practice routine of optometrists/opticians. If, in this consecutive series, an individual meets the inclusion criteria for the study, the image is uploaded to the platform. A board-certified ophthalmologist at the Medical University of Vienna then systematically checks all images individually and informs the optometrist about the need for local ophthalmologist referral.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Identification of different AMD stages on OCT images from a community-based setting to calculate the real-world prevalence of AMD | 2 years
  AMD staging will be carried out by a certified ophthalmologist at the Medical University of Vienna according to the following parameters:
  1. Healthy aging retina, including drupelets < 63 µm [3]
  2. Early AMD as defined in the protocol [3] (see 7.3 disease definitions): Medium drusen >63 µm and >125 µm. No AMD pigmentary abnormalities.
  3. Intermediate AMD as defined in the protocol [3] (see 7.3 disease definitions): Large druse > 125 µm and/or and pigmentary abnormalities
  4. Late AMD: Geographic Atrophy as defined in the protocol [3,6] (see 7.3 disease definitions)
  5. Other diseases: including neovascular AMD, RVO, DME, CCS, Stargardt disease, Pattern dystrophy, etc.

SECONDARY OUTCOMES:
Further biomarkers of AMD that are expected to be present in the cohort will be analyzed in order to assess whether they can be identified and quantified in this real-world cohort. | 2 years
  Biomarkers include:
  * Drusen presence/Refractile drusen/Hyporeflective Core Drusen (yes/no)
  * Hyperreflective foci presence (yes/no)
  * Presence of subretinal drusenoid deposits (SDD) (yes/no)
  * Loss of outer retinal layers (retinal pigment epithelium, ellipsoid zone) (scale, mm2)
  * Fluid (intraretinal fluid, subretinal fluid, pigment epithelium detachment) (yes/no)
As a post-hoc analysis, the diagnostic accuracy of AI algorithms to recognize changes associated with age-related macular degeneration in OCT volumes, will be evaluated in this real-world cohort. | 2 years